CLINICAL TRIAL: NCT02687750
Title: Testing of Radiofrequency Coil for Clinical 19F MRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Paula Foster, Professor, Western University, Canada
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RRI-PF-001
Record Dates: First submitted 2016-02-02; First posted 2016-02-22 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-02

CONDITIONS: Diagnostic Imaging

ARMS (1):
- MRI (Experimental): Eppendorf tubes containing 10% fluorine-19 diluted in agar were taped to the upper thigh of participants. Investigational device was used to image the phantom with Magnetic resonance imaging (MRI). Imaging was performed for anatomical (proton) and fluorine (agent detection). Total scan time was under 1 hour.
  Objectives:
  * Verify RF coil functionality
  * Obtain preliminary detection threshold limits using a human coil loading
  Interventions: Device: MRI

INTERVENTIONS:
Device: MRI — Investigational device is a dual tuned (fluorine/proton) MRI surface coil designed and produced by Clinical MR solutions

SUMMARY:
Testing of a dual tuned proton/fluorine MRI radio frequency coil

Images were collected from plastic fluorine phantoms taped to the upper thigh of health volunteers.

This trial was performed as part of an application for a Health Canada Investigational Device Exemption (Protocol # 226949)

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteer

Exclusion Criteria:

* MRI incompatible patient
* claustrophobia

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Verify radio frequency coil imaging functionality on humans | 1 hour of scanning
  Proof of successful MRI signal acquisition with use of investigation device.
Measure signal repeatability in different patients | 1 hour of scanning
  MRI signal strength is expected to vary slightly based on patient weight.